CLINICAL TRIAL: NCT05957523
Title: Effects of Remote Ischemic Preconditioning on Peripheral Blood Biomarkers in Healthy Adults (EMINENT): a Single-centre, Open-label, Randomized Controlled Clinical Trial
Brief Title: Effects of Remote Ischemic Preconditioning on Peripheral Blood Biomarkers in Healthy Adults (EMINENT)
Acronym: EMINENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSYY-428-02
Record Dates: First submitted 2023-06-27; First posted 2023-07-24 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Preconditioning
Keywords: Remote ischemic preconditioning; Peripheral blood; Healthy adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (high-frequency group ) (Experimental): Subjects aged 18 to 45 years and in good health agree to participate in the clinical trial and sign an informed consent form. The high-frequency remote ischemic preconditioning (RIPC) group will undergo RIPC training continuously for seven days, twice daily, with each session consisting of four cycles of 5 minutes of ischemia followed by 5 minutes of reperfusion.
  Interventions: Device: Remote ischaemic preconditioning
- Group B (low-frequency group ) (Experimental): Subjects aged 18 to 45 years and in good health agree to participate in the clinical trial and sign an informed consent form. The low-frequency RIPC group will follow the same cycle and compression pattern but will train only once a day.
  Interventions: Device: Remote ischaemic preconditioning

INTERVENTIONS:
Device: Remote ischaemic preconditioning — The participants rested in the supine position for 5 minutes, then turn on the ischaemic preconditioning apparatus and place the automatically programmed blood pressure cuff on both upper arms of the participant, pressurize to 200 mmHg, pressurize for 5 minutes, rest for 5 minutes, perform 4 cycles for a total of 40 minutes each time. The training for participants in group A will be performed once daily, while for participants in group B the training will be performed twice daily. And heart rate and blood pressure before and after each training will be recorded for 7 days.

SUMMARY:
The aim of this study is to investigate the effects of remote ischaemic preconditioning on the peripheral blood characteristics of healthy adults and to explore the possible mechanisms for improving ischaemia/reperfusion injury and its protective effects on the cardiovascular system.

DETAILED DESCRIPTION:
This study plans to recruit 60 healthy volunteers, who will be randomly divided into a high-frequency group and a low-frequency group. The high-frequency remote ischemic preconditioning (RIPC) group will undergo RIPC training continuously for seven days, twice daily, with each session consisting of four cycles of 5 minutes of ischemia followed by 5 minutes of reperfusion. The low-frequency RIPC group will follow the same cycle and compression pattern but will train only once a day. Biological samples and physiological indicators will be collected from participants on the day just before the start of ischemic preconditioning training, as well as on the 7th and 14th days following the start of the training. These samples will be analyzed to identify the differences in blood components between groups and at different time points before and after RIPC. The study aims to investigate the effects of different training frequencies of RIPC on the characteristics of peripheral blood in healthy adults, as well as the changes in the peripheral blood characteristics of the participants before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years;
* Be in good health;
* Consent to participate in the clinical trial and sign the informed consent form.

Exclusion Criteria:

* Abnormal results in biochemical checks and physiological indicators.
* Cardiovascular and cerebrovascular diseases: hypertension, coronary heart disease, congenital heart disease, cerebrovascular alterations, etc.
* Endocrine diseases: diabetes, thyroid disorders, etc.
* Hematologic diseases: anemia, paroxysmal hemoglobinuria, primary thrombocytosis, etc.
* Infectious diseases: hepatitis B, hepatitis C, syphilis, etc.
* Cancer.
* Neurological and psychiatric disorders.
* Vascular diseases: peripheral vascular disease, Raynaud's syndrome, thromboembolic diseases.
* Major trauma or surgery within the last six months.
* Pregnant or breastfeeding women.
* Upper limbs unsuitable for compression treatment: history of upper limb surgery, presence of tissue damage and limb deformity, and concomitant hemorrhagic diseases.
* Recent circumstances that may affect results: blood donors within the last month, any medication taken within the last month, fever within the last week, women within their menstrual cycle or within 7 days before the start of menstruation.
* Patients who refuse to sign the informed consent form for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in various biomarkers between intermediate and intense training group | Baseline (before training), the end of the training day (7th day from the start of training), 7th day after the end of training
  Difference in collected materials from participants in group A (intermediate RIPC training, once a day) or B (intense RIPC training, twice a day)
Change of peripheral blood characteristics | Baseline (before training), the end of the training day (7th day from the start of training), 7th day after the end of training
  Peripheral blood characteristics at different remote ischemic preconditioning, training time points, including different fractions and their characteristics expressed by the results of blood tests.
Change of gut microbiome components at different remote ischemic preconditioning training time points | Baseline (before training), the end of the training day (7th day from the start of training), 7th day after the end of training
  Gut microbiome components

SECONDARY OUTCOMES:
Incidence of adverse events | During day 1 to 7 of training.
  Incidence of adverse events related to remote ischemic preconditioning training. The adverse events were decided according to the medical records.
Change of faecal characteristics | Baseline (before training), the end of the training day (7th day from the start of training), 7rd day after the end of training
  Effect of RIPC training on faecal characteristics, expressed by the fecal test results.
Change of blood pressure | Baseline (before training), during the training session (day1-7), 7th day after the end of training.
  Changes in blood pressure at different remote ischemic preconditioning training time points, measured with sphygmomanometer.
Change of heart rates | Baseline (before training), during the training session (day1-7), 7th day after the end of training
  Changes in heart rates at different remote ischemic preconditioning training time points, measured with stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No